CLINICAL TRIAL: NCT05011240
Title: A Randomized Controlled Trial of Parent-mediated Social-communication Therapy for Young Children at Risk for Neurodevelopmental Difficulties Living in Poverty in Brazil
Brief Title: Parent-mediated Social-communication Therapy for Young Children Living in Poverty in Brazil
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Faculdade de Medicina do ABC (Other)
Responsible Party: Principal Investigator, Alicia Matijasevich, Associate Professor in Preventative Medicine, Faculdade de Medicina do ABC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 45672321.0.0000.0068
Record Dates: First submitted 2021-08-16; First posted 2021-08-18 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Child Development; Communication, Social; Environmental Exposure
Keywords: Preventative intervention; Early child development; Social communication development; Socioeconomic disadvantage; Randomized Controlled Trial
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study will be single-blinded with the researchers conducting and coding the outcome measures unaware of the intervention/control status of the study participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paediatric Autism Communication Therapy (PACT) Intervention plus Community Assistance as Usual (Experimental): Participants will receive 12 sessions over 5 months of Paediatric Autism Communication Therapy (PACT).
  Interventions: Behavioral: Paediatric Autism Communication Therapy (PACT)
- Community support as usual plus psychoeducation (Control) (Active Comparator): Participants in the Control group will receive psycho-educational support via monthly sessions led by researchers with experience in child development. In each session, a presentation will be delivered to provide parents with information about child development and environmental factors that contribute to healthy child development, including sensitive parenting styles, frequent positive social interactions between parents and children and cognitive stimulation. The presentations will be followed by group discussions. Children will also continue to receive Community Assistance as Usual via their normal early education centers. These centers offer daily activities designed to promote children's learning, autonomy, movement, integration and socialization. Children attend their educational center five days per week between the hours of 8am and 5pm.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Paediatric Autism Communication Therapy (PACT) — PACT is a parent-mediated therapy that aims to improve children's social-communication development. During PACT, a therapist uses video-feedback of parent-child play interactions to coach the parent in how to improve their sensitivity and responsiveness to their child's social-communication and interaction behaviours and to implement evidence-based strategies that facilitate social-communication development.
  Arms: Paediatric Autism Communication Therapy (PACT) Intervention plus Community Assistance as Usual
Behavioral: Psychoeducation — Control participants will receive monthly psychoeducation sessions led by a developmental specialist
  Arms: Community support as usual plus psychoeducation (Control)

SUMMARY:
Exposure to adverse environments such as socioeconomic disadvantage and psychosocial deprivation are risk-factors for neurodevelopmental problems in childhood. Children exposed to such environments may benefit from interventions that target social-communication abilities, since these skills act as protective factors for healthy neurodevelopment in vulnerable children. One early childhood intervention that has shown efficacy in improving early social-communication development is Paediatric Autism Communication Therapy (PACT). However, there are no studies testing the efficacy of PACT in Latin American countries where environmental risk factors are common. This randomized controlled trial will test the efficacy of PACT in improving social-communication development in young children at risk for neurodevelopmental difficulties due to living in socio-economically disadvantaged regions of São Paulo, Brazil.

Methods: Participants will be 160 children aged 2 years 0 months to 4 years 11 months with low social-communication abilities and their primary caregivers. Child-caregiver dyads will be recruited from public early childhood education centers in impoverished urban regions of the city of São Paulo, Brazil. Low social-communication abilities will be defined by Standard Scores <84 on the Socialization and/or Communication domains of the Vineland Adaptive Behavior Scales. Child-caregiver dyads will be randomized to receive 12 sessions (five months) of the PACT intervention (N=80) or five months of community support as usual plus psychoeducation (N=80). The primary outcome (parent-child interaction) and secondary outcomes (social-communication abilities assessed with the Vineland, neurophysiological activity during a live social interaction) will be measured pre- and post-intervention. All procedures will be performed in accordance with the CONSORT declaration for non-pharmacological interventions.

ELIGIBILITY:
Inclusion Criteria:

* aged 2 years 0 months to 4 years 11 months
* low social-communication abilities indexed by Standardized Scores between 55 to 84 on the Socialization and/or Communication Domains of the Vineland Adaptive Behavior Scales - Third Edition
* parent/primary caregiver agrees to participate in the trial

Exclusion Criteria:

* known neurological condition such as epilepsy
* known genetic disorder such as Down Syndrome
* hearing or visual impairment in the parent or child that could interfere with the intervention
* self-reported current psychiatric or neurological disorder in the parent that could interfere with the intervention

Ages: 24 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in parent-child interaction synchrony | Change from baseline (week 1, pre-intervention) to 5 month (post-intervention)
  Parent-child interaction synchrony will be measured during a 10-minute free-play interaction between the primary caregiver and child and coded using the Dyadic Communication Measure for Autism (DCMA). Synchrony is coded as the proportion of communicative behaviors of the primary caregiver that elicit responses from the child.

SECONDARY OUTCOMES:
Change in Socialization and Communication Domain Standardized Scores on the Vineland Adaptive Behavior Scales - 3 | Change from baseline (week 1, pre-intervention) to 5 month (post-intervention)
  Parent-reported measure of children's adaptive social and communication skills
Change in neurophysiological activity during live social interaction | Change from baseline (week 1, pre-intervention) to 5 month (post-intervention)
  Neurophysiological activity measured with electroencephalography (EEG) during a live play interaction between the child and an examiner
Change in Internalizing and Externalizing Behavior Problems | Change from baseline (week 1, pre-intervention) to 5 month (post-intervention)
  Internalizing and externalizing behaviour problems measured by parent-report on the Child Behavior Checklist 1.5-5 and on the Strengths and Difficulties Questionnaire 2-4.
Child initiations during parent-child interaction | Change from baseline (week 1, pre-intervention) to 5 month (post-intervention)
  Child initiations will be measured during a 10-minute free-play interaction between the primary caregiver and child and coded using the Dyadic Communication Measure for Autism (DCMA). Child initiations are coded as the proportion of the child's spontaneous communicative behaviors oriented to the parent, including verbal and non-verbal behaviors.

OTHER OUTCOMES:
Change in style of parenting care | Change from baseline (week 1, pre-intervention) to 5 month (post-intervention)
  Self-reported parenting care style measured by the Parenting Scale
Change in parent-child joint engagement | Change from baseline (week 1, pre-intervention) to 5 month (post-intervention)
  Joint interaction behaviors between parent and child during free-play interaction measured with the Joint Engagement Rating Inventory
Change in developmental ability | Change from baseline (week 1, pre-intervention) to 5 month (post-intervention)
  Global developmental ability measured by the Ages and Stages Questionnaire completed by primary caregivers.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Godoy PBG, Shephard E, Argeu A, Silveira LR, Salomone E, Aldred C, Green J, Polanczyk GV, Matijasevich A. Social communication therapy for children at risk for neurodevelopmental difficulties: Protocol for a clinical trial. Ann N Y Acad Sci. 2022 Aug;1514(1):104-115. doi: 10.1111/nyas.14784. Epub 2022 May 4. PMID 35506888